CLINICAL TRIAL: NCT01744041
Title: Perinatal Depression: Dyadic-IPT to Improve Health of Mother and Baby
Brief Title: Mommy-Baby Treatment for Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201203136; K23MH090245 (NIH)
Record Dates: First submitted 2012-11-27; First posted 2012-12-06 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Depressive Disorder, Major; Postpartum Depression
Keywords: depression; pregnancy; postpartum; psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression, Postpartum; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dyadic Interpersonal Psychotherapy (Experimental): Brief Interpersonal Psychotherapy during pregnancy followed by dyadic mother-infant psychotherapy for one year postpartum
  Interventions: Behavioral: Dyadic Interpersonal Psychotherapy
- Enhanced Treatment as Usual (Active Comparator): Personalized referral to community resources for depression treatment
  Interventions: Other: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: Dyadic Interpersonal Psychotherapy — This intervention consists of a brief psychotherapeutic intervention, Interpersonal Psychotherapy, during pregnancy. Interpersonal Psychotherapy focuses on improving social relationships and interpersonal communication to improve mood. The postpartum phase also utilizes developmentally appropriate strategies to improve the mother-infant relationship.
  Arms: Dyadic Interpersonal Psychotherapy
Other: Enhanced Treatment as Usual — This intervention consists of personalized referrals to specialty mental health providers, spiritual counselors, or other needed social services. It includes some non-specific supportive techniques delivered primarily via telephone.
  Arms: Enhanced Treatment as Usual

SUMMARY:
Perinatal depression is a major public health problem, affecting 15% of women during pregnancy through the postpartum period, with adverse consequences for the mother, the fetus, the infant, and the family. Despite increasing evidence of the importance of this critical risk interval, little research has investigated the effects of depression treatment during pregnancy on infant outcomes. The purpose of this study is to test the feasibility, acceptability, and effectiveness of a new intervention, Interpersonal psychotherapy for the mother-infant dyad (IPT-Dyad). This intervention begins during pregnancy and continues with the mother and infant until one year postpartum. The investigators hypothesize that IPT-Dyad will be better than treatment as usual in reducing depressive symptoms, improving psychosocial functioning,increasing parenting self-efficacy, improving infant emotional development, and enhancing mother-infant relationship quality.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 18 years and older
* between 12 and 30 weeks gestation
* Score greater than or equal to 13 on Edinburgh Depression Scale
* Structured Clinical Interview (SCID-IV) diagnosis of Major Depressive Disorder, dysthymia, or Depressive Disorder, Not otherwise Specified
* English Speaking

Exclusion Criteria:

* Substance abuse or dependence in past 3 months
* Active suicidal or homicidal ideation
* Bipolar disorder, psychotic disorder
* unstable medical condition or other medical/obstetrical complication
* Evidence of severe intimate partner violence
* Ongoing psychosocial or pharmacotherapy for depression

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-11; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Lenze, Ph.D., Principal Investigator — Washington Univeristy
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Lenze SN, Rodgers J, Luby J. A pilot, exploratory report on dyadic interpersonal psychotherapy for perinatal depression. Arch Womens Ment Health. 2015 Jun;18(3):485-91. doi: 10.1007/s00737-015-0503-6. Epub 2015 Jan 22. PMID 25604869
- [Result] Lenze SN, Potts MA. Brief Interpersonal Psychotherapy for depression during pregnancy in a low-income population: A randomized controlled trial. J Affect Disord. 2017 Mar 1;210:151-157. doi: 10.1016/j.jad.2016.12.029. Epub 2016 Dec 20. PMID 28038377
- [Derived] Lenze SN, Potts MA, Rodgers J, Luby J. Lessons learned from a pilot randomized controlled trial of dyadic interpersonal psychotherapy for perinatal depression in a low-income population. J Affect Disord. 2020 Jun 15;271:286-292. doi: 10.1016/j.jad.2020.03.084. Epub 2020 Apr 15. PMID 32479328

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dyadic Interpersonal Psychotherapy | Enhanced Treatment as Usual
Started | 21 | 21
Completed | 15 | 13
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dyadic Interpersonal Psychotherapy | Enhanced Treatment as Usual | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (5.81) | 26.38 (5.9) | 26.64 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 16 | 33
  White | 4 | 3 | 7
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42
Edinburgh Depression Scale score [Mean (Standard Deviation); unit: units on a scale] — 10-item scale, total score reported, minimum score is 0 and maximum score is 30, higher scores indicate worse outcome
  units on a scale | 17.81 (3.71) | 17.90 (4.60) | 17.86 (4.13)

OUTCOME MEASURES:

1. Primary Outcome: Change in Edinburgh Depression Scale From Baseline
Description: Edinburgh Postnatal Depression Scale, a 10-item scale of depression severity, scores range from 0 to 30 with higher scores indicating worse outcome.
Time Frame: Change from baseline at End of pregnancy (between 37-39 weeks gestation); change from baseline at 3 months postpartum; change from baseline at 6 months postpartum; change from baseline at 9 months postpartum; change from baseline at 12 months postpartum
Population: Data shown are for the participants who completed study questionnaires at that time-point. Due to participant drop-out, this number may be less than the overall number of participants analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dyadic Interpersonal Psychotherapy | Enhanced Treatment as Usual
Number analyzed (Participants) | 21 | 21
units on a scale
  Baseline Score | 17.81 (3.71) | 17.9 (4.6)
  37-39 week gestation score | 12.04 (1.22) | 11.41 (1.72)
  3-month postpartum score: number analyzed (Participants) | 14 | 16
  3-month postpartum score | 11.0 (6.1) | 10.3 (6.8)
  6-month postpartum score: number analyzed (Participants) | 15 | 14
  6-month postpartum score | 9.5 (2.9) | 9.4 (5.8)
  9-month postpartum score: number analyzed (Participants) | 14 | 12
  9-month postpartum score | 10.6 (5.9) | 9.4 (4.7)
  12-month postpartum score: number analyzed (Participants) | 15 | 13
  12-month postpartum score | 10.8 (4.0) | 8.8 (4.9)

ADVERSE EVENTS:
Time Frame: Baseline to 12 months postpartum, ranging from 14 to 40 months
Arm/Group | Dyadic Interpersonal Psychotherapy | Enhanced Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

LIMITATIONS AND CAVEATS:
This is a small pilot study designed to assess feasibility and not efficacy of this intervention. The primary outcome measure was a self-report scale that may not reflect unbiased outcomes. There was a substantial drop-out rate in each study arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT01744041/Prot_SAP_000.pdf